CLINICAL TRIAL: NCT04321239
Title: Feasibility of a Technology-Enabled Chronic Pain Self-Management Intervention Delivered by Community Health Workers
Brief Title: Positive Psychology for Chronic Pain Self-management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute on Aging (NIA) (NIH); Weill Medical College of Cornell University (Other)
Responsible Party: Principal Investigator, Mary Janevic, Associate Research Scientist, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUM00162275; 2P30AG022845-16 (NIH)
Record Dates: First submitted 2020-03-23; First posted 2020-03-25 (Actual); Results first posted 2021-11-01 (Actual); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Participants will engage in a 7-week positive psychology-based chronic pain self-management program.
  Interventions: Behavioral: Positive STEPS
- Usual care control group (No Intervention): After completing the follow-up telephone survey, individuals in the control condition will be given access to the online program, a wearable physical activity tracker to use and keep, and will be invited to attend a one-time 2.5-hour in-person or telephone workshop that summarizes intervention content and that will be led jointly by study staff and a community health worker.

INTERVENTIONS:
Behavioral: Positive STEPS — Individuals in the intervention group will meet with a community health worker at an in-person or virtual study orientation session. At this session, they will be introduced to the program, learn how to use the online modules and any associated materials, and choose a day and time for future weekly telephone sessions. Participants will also be given a wearable physical activity tracker at the orientation session to use throughout the course of the program. They can choose to report daily step counts either by automatically syncing to an app or by manual reporting via text message. The program will be delivered over 6 weeks. Each week participants will complete a web-based module and have one telephone session with the community health worker to discuss that module and to set a related goal. Participants will also set weekly goals related to walking, which will be informed and tracked by daily step-counts from the physical activity tracker.
  Arms: Intervention group

SUMMARY:
Learning chronic pain self-management skills can help patients improve daily functioning and quality of life, while avoiding risks associated with opioids and other pharmacological treatments. Community health workers (CHWs) may help make chronic pain self-management interventions more accessible to older adults living in underserved communities. The goal of this study is to conduct a randomized pilot and feasibility trial of a positive psychology-based chronic pain self-management intervention delivered by CHWs, in conjunction with mobile health tools, in a sample of 50 older adults recruited from community sites in Detroit, Michigan. This study will involve the use of mixed quantitative and qualitative methods to assess participant engagement and satisfaction, and change in pain-related outcomes.

ELIGIBILITY:
Inclusion Criteria:

* English-proficient
* Ambulatory with or without assistive device
* Community-living
* Have a cell or landline phone
* Have Internet access (home or elsewhere);
* Self-reported chronic musculoskeletal pain (pain in muscles or joints for > 3 months); >4 (0-10 scale) average pain level over last week; >1 day/previous 30 when pain made it difficult to do usual activities.

Exclusion Criteria:

* Serious acute illness or hospitalization in last month
* Planned surgery in next three months
* Severe cognitive impairment or other severe physical or psychiatric disorder judged by study team to pose significant barrier to deriving program benefit

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2020-05-14 (Actual); Primary Completion 2020-12-22 (Actual); Study Completion 2020-12-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary Janevic, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes
1. Self-reported survey data (baseline and 8 weeks from baseline) on pain and functioning, as well as other health and demographic information from a telephone survey of 50 pilot study participants. For 25 of these participants, we will also have up to six weeks of daily activity (step count) data. Two anonymized datasets will be created: 1) survey data only; 2) survey data plus, for the subset of 25 participants, activity data linked to survey data. In order to maintain confidentiality, outliers, dates, and personal identifiers will be removed from the data set.
  2. Notes from post-program qualitative interviews (n=25). These are in-depth, semi-structured interviews about challenges, facilitators, and satisfaction with various aspects of the program and its implementation. We will share de-identified copies of detailed notes from these interviews (we do not plan on producing verbatim transcripts) but not audiorecordings.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available for sharing upon the date of online publication of the results of the primary aims.

REFERENCES:
- [Derived] Janevic M, Robinson-Lane SG, Courser R, Brines E, Hassett AL. A Community Health Worker-Led Positive Psychology Intervention for African American Older Adults With Chronic Pain. Gerontologist. 2022 Oct 19;62(9):1369-1380. doi: 10.1093/geront/gnac010. PMID 35394525

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention Group: Participants will engage in a 7-week positive psychology-based chronic pain self-management program.
  Positive STEPS: Individuals in the intervention group will meet with a community health worker at an in-person or virtual study orientation session. At this session, they will be introduced to the program, learn how to use the online modules and any associated materials, and choose a day and time for future weekly telephone sessions. Participants will also be given a wearable physical activity tracker at the orientation session to use throughout the course of the program. They will report daily step counts via text message. The program will be delivered over 6 weeks. Each week participants will complete a web-based module and have one telephone session with the community health worker to discuss that module and to set a related goal. Participants may also set weekly goals related to walking, which will be informed and tracked by daily step-counts from the physical activity tracker.
Period: Overall Study
Arm/Group | Intervention Group | Usual Care Control Group
Started | 25 | 26
Completed | 22 | 24
Not Completed | 3 | 2

BASELINE CHARACTERISTICS:
Population: All participants who were randomized to a treatment condition and completed baseline survey.
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Group | Usual Care Control Group | Total
Number analyzed (Participants) | 25 | 26 | 51
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: age data not available for one participant
  years
    number analyzed (Participants) | 25 | 25 | 50
    (all) | 71.6 (6.7) | 71.9 (7.6) | 71.8 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 23 | 46
  Male | 2 | 3 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 25 | 25 | 50
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 23 | 24 | 47
  White | 0 | 0 | 0
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 25 | 26 | 51
Pain interference (PROMIS 6-item scale) [Mean (Standard Deviation); unit: T-score] — The Pain Interference 6-item subscale of the Patient-Reported Outcomes Measurement Information System (PROMIS)-43 Adult Profile. Items ask how much pain in the last 7 days has interfered with daily activities such as household chores and social activities (1=not at all to 5=very much); raw total scale scores range from 6 (low interference) to 30 (high interference). When converted to T-scores (normed such that a score of 50 is the population mean and 10 T-score points=1 standard deviation), the possible range is 42 to 76, with a higher score representing worse outcome. Population: Two participants had missing data on this measure.
  T-score
    number analyzed (Participants) | 23 | 26 | 49
    (all) | 59.8 (6.6) | 59.1 (7.9) | 59.4 (7.3)
Physical functioning (PROMIS 4-item scale) [Mean (Standard Deviation); unit: T-score] — The Physical Functioning 4-item subscale of the Patient-Reported Outcomes Measurement Information System (PROMIS)-29 Adult Profile. Items ask how much difficulty participant has in doing daily activities such as household chores, using stairs, and walking 15 minutes (1=without any difficulty to 5=unable to do); raw total scale scores range from 4 (high functioning) to 20 (low functioning). When converted to T-scores (normed such that a score of 50 is the population mean and 10 T-score points=1 standard deviation), the possible range is 23 to 57, with a higher score representing worse outcome.
  T-score | 41.1 (7.0) | 40.8 (6.4) | 40.9 (6.7)
Social participation (PROMIS 4-item scale) [Mean (Standard Deviation); unit: T-score] — Ability to Participate in Social Roles and Activities, a 4-item subscale from PROMIS-20 rating the amount of trouble (1=not at all to 5=very much) in participating in social roles such as family activities, leisure activities, and work. Raw total scale scores range from 4 (high functioning) to 20 (low functioning). When converted to T-scores (normed such that a score of 50 is the population mean and 10 T-score points=1 standard deviation), the possible range is 29 to 64, with a higher score representing worse outcome. Population: Missing data (missing items) on this measure for a total of 4 participants.
  T-score
    number analyzed (Participants) | 23 | 24 | 47
    (all) | 49.4 (9.4) | 48.2 (8.9) | 48.8 (9.1)
Resilience (Connor-Davidson 10-item scale) [Mean (Standard Deviation); unit: units on a scale] — 10-item version of the Connor-Davidson resilience scale rating the degree (0=not true at all to 4=true nearly all the time) respondent can cope/be resilient in various situations. Higher score means more resilience.
  units on a scale | 3.1 (0.56) | 3.3 (0.49) | 3.2 (0.52)
Pain Self-Efficacy [Mean (Standard Deviation); unit: units on a scale] — The Pain Self-Efficacy Questionnaire, a 10-item scale (Nicholas 1989) rating confidence at doing specific things (e.g., chores, accomplishing goals, becoming more active) despite pain; each item scored from 0=not at all confident to 6=completely confident.
  units on a scale | 4.7 (1.3) | 4.4 (1.3) | 4.5 (1.3)
Pain intensity (0 to 10) [Mean (Standard Deviation); unit: units on a scale] — A numeric rating scale ranging from 0 (no pain at all; best outcome) to 10 (worst pain you can imagine; worst outcome)
  units on a scale | 6.3 (1.9) | 6.4 (1.5) | 6.4 (1.7)

OUTCOME MEASURES:

1. Primary Outcome: Change in Pain Interference
Description: The Pain Interference 6-item subscale of the Patient-Reported Outcomes Measurement Information System (PROMIS)-43 Adult Profile. Items ask how much pain in the last 7 days has interfered with daily activities such as household chores and social activities (1=not at all to 5=very much); raw total scale scores range from 6 (low interference) to 30 (high interference). When converted to T-scores (normed such that a score of 50 is the population mean and 10 T-score points=1 standard deviation), the possible range is 42 to 76, with a higher score representing worse outcome.
Time Frame: Baseline and 8 weeks
Population: Participants who had data on both baseline and follow-up measure. Change score is the follow-up minus baseline score, such that a greater, negative change value is a better outcome.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Intervention Group | Usual Care Control Group
Number analyzed (Participants) | 21 | 23
T-score | -3.82 (5.2) | .32 (5.0)

2. Primary Outcome: Change in Self-reported Physical Functioning
Description: The Physical Functioning 4-item subscale of the Patient-Reported Outcomes Measurement Information System (PROMIS)-29 Adult Profile. Items ask how much difficulty participant has in doing daily activities such as household chores, using stairs, and walking 15 minutes (1=without any difficulty to 5=unable to do); raw total scale scores range from 4 (high functioning) to 20 (low functioning). When converted to T-scores (normed such that a score of 50 is the population mean and 10 T-score points=1 standard deviation), the possible range is 23 to 57, with a higher score representing worse outcome.
Time Frame: Baseline and 8 weeks
Population: Participants who had both baseline and follow-up data on this measure.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Intervention Group | Usual Care Control Group
Number analyzed (Participants) | 22 | 24
T-score | 43.7 (7.7) | 40.9 (6.3)

3. Secondary Outcome: Participant Global Impression of Change--Pain
Description: How participant thinks their pain has changed from baseline (much worse (1) to much better (7)). Higher score represents a better outcome.
Time Frame: Baseline and 8 weeks
Population: Participants with baseline and follow-up data on this measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention Group | Usual Care Control Group
Number analyzed (Participants) | 21 | 24
units on a scale | 6.1 (.97) | 4.4 (1.3)

4. Secondary Outcome: Change in Pain Self-efficacy
Description: The Pain Self-Efficacy Questionnaire, a 10-item scale (Nicholas 1989) rating confidence at doing specific things (e.g., chores, accomplishing goals, becoming more active) despite pain; each item scored from 0=not at all confident to 6=completely confident.
Time Frame: Baseline and 8 weeks
Population: Participants who had data on both baseline and follow-up measure. Change score is the follow-up minus baseline score, such that a greater, positive change value is a better outcome.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention Group | Usual Care Control Group
Number analyzed (Participants) | 22 | 24
units on a scale | .36 (.91) | -.16 (.71)

5. Secondary Outcome: Change in Social Participation
Description: Ability to Participate in Social Roles and Activities, a 4-item subscale from PROMIS-20 rating the amount of trouble (1=not at all to 5=very much) in participating in social roles such as family activities, leisure activities, and work. Raw total scale scores range from 4 (high functioning) to 20 (low functioning). When converted to T-scores (normed such that a score of 50 is the population mean and 10 T-score points=1 standard deviation), the possible range is 29 to 64, with a higher score representing worse outcome.
Time Frame: Baseline and 8 weeks
Population: Participants who had data on both baseline and follow-up measure. Change score is the follow-up minus baseline score, such that a greater, negative change value (or smaller positive change) is a better outcome.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Intervention Group | Usual Care Control Group
Number analyzed (Participants) | 18 | 23
T-score | .11 (4.4) | .17 (3.3)

6. Secondary Outcome: Change in Resilience
Description: 10-item version of the Connor-Davidson resilience scale rating the degree (0=not true at all to 4=true nearly all the time) respondent can cope/be resilient in various situations. Higher score means more resilience.
Time Frame: Baseline and 8 weeks
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention Group | Usual Care Control Group
Number analyzed (Participants) | 21 | 24
units on a scale | .10 (.38) | -.02 (.44)

7. Secondary Outcome: Participant Global Impression of Change - Functioning
Description: How participant thinks their functioning has changed from baseline (much worse (1) to much better (7)). Higher score represents a better outcome.
Time Frame: 8 weeks
Population: Participants with baseline and follow-up data on this measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention Group | Usual Care Control Group
Number analyzed (Participants) | 21 | 24
units on a scale | 6.4 (.74) | 4.6 (1.4)

ADVERSE EVENTS:
Time Frame: Two months
Arm/Group | Intervention Group | Usual Care Control Group
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/26
Serious Adverse Events (participants affected / at risk) | 2/25 | 0/26
Other Adverse Events (participants affected / at risk) | 0/25 | 0/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intervention Group (N=25) | Usual Care Control Group (N=26)
hospitalization (Musculoskeletal and connective tissue disorders) | 1 | 0 — Participant had a fall; was determined to be unrelated to the intervention.
hospitalization (Cardiac disorders) | 1 | 0 — Participant hospitalized with chest pain; determined to be unrelated to intervention.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-07-01): https://cdn.clinicaltrials.gov/large-docs/39/NCT04321239/Prot_SAP_000.pdf
  • Informed Consent Form (2020-07-01): https://cdn.clinicaltrials.gov/large-docs/39/NCT04321239/ICF_001.pdf